CLINICAL TRIAL: NCT07249333
Title: Effect of Neoadjuvant Radiotherapy on the Incidence of Perioperative Complications After Radical Surgical Treatment of Colorectal Cancer
Brief Title: Perioperative Complications After Neoadjuvant Radiotherapy for Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Vojvodina (Other Government)
Responsible Party: Principal Investigator, Nora Mihalek, Asist. Dr., Oncology Institute of Vojvodina
Other Study IDs: 4/25/1-2086/2-2
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Neoadjuvant Radiotherapy; Perioperative Complication
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant radiotherapy group: Patients who underwent radiotherapy before the surgical treatment of colorectal cancer
- Control group: Patients who did not undergo radiotherapy before the surgical treatment of colorectal cancer

SUMMARY:
Neoadjuvant radiotherapy plays an important role in the treatment of locally advanced colorectal cancer. Although radiation therapy is extremely important in reducing the tumor mass, downstaging, and therefore providing conditions for curative surgery, neoadjuvant therapy can increase the risk of perioperative complications, which can lead to slower patient recovery, greater perioperative morbidity, prolonged hospitalization, and increased treatment costs.

The aim of the study is to determine whether there is a difference in the incidence of perioperative complications after radical colorectal cancer surgery between patients who received neoadjuvant radiotherapy and those patients who did not undergo neoadjuvant radiation.

Data is collected from the medical documentation and information system of the Oncology Institute of Vojvodina. Demographic characteristics of patients, comorbidities, length of hospital stay, length of treatment in the intensive care unit, occurrence of complications in the perioperative period, as well as data on neoadjuvant therapy are analyzed. All included patients are of similar general condition, as determined by the CFS (Clinical Frailty Scale). Intraoperative complications are graded using the ClassIntra classification of intraoperative adverse events, and the presence of postoperative adverse events are assessed and classified using the Clavien-Dindo classification of postoperative complications and the HARM (HospitAl stay, Readmission, Mortality rate) score.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years of age)
* Clinical Frailty Scale 2, 3 or 4 status
* Patients undergoing radical surgical treatment of colorectal cancer

Exclusion Criteria:

* Patients undergoing palliative surgical treatment of colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective radical colorectal cancer surgery in the period between 01.06.2024. and 30.06.2026. in the Oncology Institute of Vojvodina.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of particular perioperative complications (surgical site infection, urinary infection, wound dehiscence, bowel anastomosis dehiscence, ileus, reoperation) | During hospital stay (assessed up to 15 days)
  Data collected from medical records and information system

SECONDARY OUTCOMES:
ClassIntra classification of intraoperative adverse events | Perioperative/Periprocedural
  Maximal value: 5; Minimal value: 0 (higher score indicates worse outcome)
Clavien-Dindo classification of postoperative adverse events | During hospital stay (assessed up to 15 days)
  Maximal value: 5; Minimal value: 1 (higher score indicates worse outcome)
HARM (Hospital stay, Readmission, Mortality) scale of postoperative adverse events | During hospital stay (assessed up to 15 days)
  Maximal value: 5; Minimal value: 0 (higher score indicates worse outcome)
Length of hospital stay | During hospital stay (assessed up to 15 days)
  Number of days spent in hospital
Length of intensive care unit stay | During hospital stay (assessed up to 15 days)
  Number of days spent in the intensive care unit
Duration of antibiotic use (Days of Therapy - DOT) | During hospital stay (assessed up to 15 days)
  Number of days when antibiotic therapy was applied. In the case of multiple antibiotic administration, each antibiotic is counted separately and DOT is the sum of each antibiotic therapy duration in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Vojvodina, Kamenitz, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No